CLINICAL TRIAL: NCT06731153
Title: A Randomized, Controlled, Open-label, Phase II Clinical Study Evaluating the JAK1 Inhibitor Ivarmacitinib to Reverse Immunotherapy Resistance in Triple-negative Breast Cancer
Brief Title: JAK1 Inhibitor Ivarmacitinib Reversing Immunotherapy Resistance in TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N085
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Triple Negative Breast Cancer (TNBC); Metastatic Breast Cancer
Keywords: immune resistance; JAK1 inhibitor; triple negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — ivarmacitinib; camrelizumab; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety run-in (Experimental): Ivarmacitinib + Camrelizumab + Eribulin
  Interventions: Drug: Ivarmacitinib; Drug: Camrelizumab (SHR-1210); Drug: Eribulin
- Treatment group (Experimental): Ivarmacitinib + Camrelizumab + Eribulin, RP2D
  Interventions: Drug: Ivarmacitinib; Drug: Camrelizumab (SHR-1210); Drug: Eribulin
- Control group (Active Comparator): Ivarmacitinib + Eribulin, RP2D
  Interventions: Drug: Ivarmacitinib; Drug: Eribulin

INTERVENTIONS:
Drug: Ivarmacitinib — a selective Janus kinase 1 inhibitor
Drug: Camrelizumab (SHR-1210) — a humanised anti-programmed death-1 (anti PD-1) antibody
  Arms: Safety run-in; Treatment group
Drug: Eribulin — Eribulin is an anticancer drug approved for treatment of metastatic breast cancer. This drug is a synthetic derivative from Japanese marine sponge Halichondria okadai. It acts by interfering with the microtubular growth ultimately leading to apoptosis after prolonged mitotic blockage.

SUMMARY:
This is a prospective, open-label, randomized phase II clinical study which recruits unresectable recurrent or metastatic triple-negative breast cancer resistant to immunotherapy.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized phase II clinical study. The purpose of this study is to test the combination of the JAK1 inhibitor Ivarmacitinib and the PD-1 inhibitor Camrelizumab in patients with immunotherapy-resistant locally advanced inoperable or metastatic triple-negative breast cancer. The study included a safety run-in period to explore the safety of Ivarmacitinib in combination with Eribulin and Camrelizumab, which will provide a recommended dose for the triplet combination of Ivarmacitinib, Camrelizumab and Eribulin. The latter phase II period is set to compare the efficacy of the triplet combination of Ivarmacitinib, Camrelizumab and Eribulin versus Eribulin plus Ivarmacitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old (both ends included);
2. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0,1, 2;
3. Metastatic or locally advanced, histologically documented TNBC;
4. Histologically confirmed diagnosis of TNBC characterized by estrogen-receptor negative (ER-), progesterone receptor negative (PR-) and human epidermal growth factor-2 receptor negative (HER2-);
5. Radiologic/objective evidence of recurrence or disease progression after immunotherapy (anti-PD-1/PD-L1 antibodies) for metastatic breast cancer (MBC);
6. For patients refractory/resistant to anti-PD-1/PD-L1 antibodies, there should be no anti-PD-1/PD-L1 treatment-related toxicity from prior therapies;
7. Participants must have measurable disease per RECIST 1.1;
8. Life expectancy ≥3 months;
9. The functions of the main organs are basically normal and meet the following conditions:

   I. Blood routine examination criteria shall meet: HB ≥90 g/L (no blood transfusion within 14 days); The ANC acuity 1.5 x 10^9 / L; PLT acuity 90 x 10^9 / L; II. Biochemical tests should meet the following criteria: Albumin ≥3.0 g/dL; TBIL≤1.5×ULN (upper limit of normal value); ALT and AST ≤3×ULN; If liver metastases were present, ALT and AST≤ 5×ULN; Serum Cr ≤1.5×ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula); International Normalized ratio (INR)≤ 1.5 or prothrombin time ≤1.5 times ULN; Activated partial thromboplastin time (aPTT)≤1.5 times ULN III. Male QTcF ≤450 msec, female QTcF ≤470 msec; LVEF≥50%;
10. They have not received radiotherapy, molecular targeted therapy, or surgery within 3 weeks before the start of the study, and have recovered from the acute toxicity of previous treatment (if surgery was performed, the wound has healed completely); No peripheral neuropathy or grade I peripheral neurotoxicity;
11. Fertile female subjects were required to use a medically approved contraceptive method during the study treatment period and for at least 3 months after the last use of the study drug;
12. Subjects volunteered to join the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Active brain metastases, cancerous meningitis, primary central nervous system (CNS) tumors not treated with surgery or radiotherapy; Stable for at least 4 weeks after treatment and corticosteroid discontinuation >2 weeks can be included;
2. History of active autoimmune disease or autoimmune disease that may recur (excluding well-controlled type 1 diabetes, hypothyroidism (which can be controlled with hormone replacement therapy only), well-controlled celiac disease, skin diseases that do not require systemic treatment (e.g. Vitiligo, psoriasis, alopecia) , any other disease that is not expected to recur without an external trigger);
3. Have previously received Eribulin;
4. Any active malignancies ≤2 years prior to first administration of the drug, except for the specific cancers studied in this trial and any locally recurrent cancers that have been treated with radical treatment (such as resected basal cell or squamous cell skin cancer, cervical or breast carcinoma in situ);
5. Have an active autoimmune disease, or a disease requiring systemic steroid hormone or immunosuppressive drug treatment, or other acquired (HIV infection), congenital immunodeficiency disease, or a history of organ transplantation (including allogeneic bone marrow transplantation);
6. Corticosteroids ≤14 days before the first administration of the study drug;
7. Uncontrolled diabetes mellitus, ≥grade 3 hypoalbuminemia, or laboratory tests were present ≤14 days before the first administration of the study drug or >Grade 1 abnormalities in blood potassium, sodium, or calcium despite standard drug therapy;
8. History of interstitial lung disease, non-infectious pneumonia, or uncontrolled disease, including pulmonary fibrosis and acute lung disease;
9. Severe chronic or active infections (including tuberculosis, etc.) requiring systemic antimicrobial, antifungal, or antiviral therapy within 14 days prior to the first administration of the drug. Note: Antiviral therapy is allowed for patients with viral hepatitis
10. Active psychiatric disorders (schizophrenia, major depressive disorder, bipolar disorder, etc.). Depression being treated with antidepressants is not an exclusion criterion;
11. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA > 500 IU/mL) or active HCV carriers with detectable HCV RNA. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL) can be enrolled;
12. Any major surgery requiring general anesthesia ≤28 days before the first administration of the drug;
13. Previous allogeneic stem cell transplantation or organ transplantation;
14. Any of the following cardiovascular criteria

    1. The presence of cardiogenic chest pain ≤28 days
    2. The presence of symptomatic pulmonary embolism ≤28 days
    3. To investigate any history of acute myocardial infarction ≤6 months
    4. A history of heart failure ≤6 months at any New York Heart Association (NYHA) grade III or IV
    5. Presence of any ventricular arrhythmia event ≤6 months of grade 2 or greater severity
    6. Any history of cerebrovascular accidents ≤6 months
    7. Corrected QT Interval (QTc)(corrected by Fridericia method) >450 ms.
15. Any syncope or seizure that occurred ≤28 days;
16. Poorly controlled hypertension (defined as: systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg)
17. Hypersensitivity to ivarmacitinib or to any component of containers;
18. Systemic chemotherapy within 28 days of initial administration of the investigational drug or immunotherapy (e.g., interleukin, interferon, thymosin, etc.), hormone therapy, targeted therapy, or any investigational therapy within 14 days of initial administration of the investigational drug or within 5 half-lives, whichever is shorter;
19. Use of any Chinese herbal medicine or proprietary Chinese medicine with anti-cancer activity approved by the National Drug Administration (NMPA) within 14 days prior to first administration of the investigational drug (regardless of cancer type);
20. Toxicity from previous anticancer therapy has not improved to baseline or stabilized, except for AEs not considered a safety risk (e.g., hair loss, neuropathy, and specific laboratory abnormalities);
21. Have received live vaccine ≤28 days before. Note: Seasonal influenza vaccine is an inactivated vaccine in a broad sense and is allowed to be used. Intranasal influenza vaccine is a live vaccine and should not be used;
22. An underlying medical condition (including laboratory abnormalities), alcohol or drug abuse or dependence that impedes study drug administration or interferes with interpretation of study drug toxicity and AE, or results in inadequate or reduced adherence to the study;
23. Concurrent participation in another clinical study, unless it is an observational (non-interventional) clinical study or in the follow-up period of an interventional study;
24. Inability to swallow capsules or diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, total stomach or small intestine resection, bariatric surgery, inflammatory bowel disease, or incomplete or complete intestinal obstruction;
25. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion requiring frequent drainage or medical intervention within 7 days of first administration of the drug (clinically significant recurrence requiring additional intervention within 2 weeks after intervention, excluding exudate cytological testing);
26. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety run-in: Incidence rate of dose-limiting toxicities (DLTs) | 21±3 days
  Incidence rate of DLT will be evaluated in participants in the Safety Run-In, who will be followed for protocol-defined DLT events up to 21±3 days after the first dose of Ivarmacitinib + Camrelizumab + Eribulin.
Safety run-in: adverse events (AEs) | 21±3 days
  Incidence rate of AEs of any cause will be evaluated in participants in the Safety Run-In according to CTCAE v5.0.
Safety run-in: Serious adverse events (SAEs) | 21±3 days
  Incidence rate of SAEs of any cause will be evaluated in participants in the Safety Run-In according to CTCAE v5.0.
Objective response rate (ORR) | The observation period related to this endpoint is up to 12 months.
  Defined as the proportion of patients with complete response (CR) and partial response (PR) by magnetic resonance imaging (MRI) or Computed Tomography (CT) according to RECIST v1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | The observation period related to this endpoint is up to 12 months.
  Defined as the proportion of participants with CR and PR as the best overall response.
Duration of Response (DOR) | The observation period related to this endpoint is up to 12 months.
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause). Participants without reported events are censored at the last disease evaluation.
Progression Free Survival (PFS) | The observation period related to this endpoint is up to 12 months.
  PFS based on Kaplan-Meier methodology will be defined as the time from randomization until the identification of disease progression or death, whichever occurs first. Subjects without disease progression or death at the time of analysis will be censored at the date of last disease evaluation.
Overall Survival (OS) | The observation period related to this endpoint is up to 24 months.
  Overall survival based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Treatment-Related Toxicity Rate | The observation period related to this endpoint is up to 12 months.
  The percentage of participants who experienced any grade treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No